CLINICAL TRIAL: NCT03601026
Title: Interdisciplinary Approach to Maximize Adolescent Potential: Genetic Counselling Interventions to Reduce Negative Environmental Effects
Brief Title: Genetic Counselling in the Prevention of Mental Health Consequences of Cannabis Use
Acronym: IMAGINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IMGN18
Record Dates: First submitted 2018-07-05; First posted 2018-07-26 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Mental Illness; Schizophrenia; Bipolar Disorder; Major Depressive Disorder; Cannabis Use; Psychosis
Keywords: Severe mental illness; Developmental psychopathology; Trial-within-cohort; Genetic counselling; Cannabis use; Prevention
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Bipolar Disorder; Depressive Disorder, Major; Psychotic Disorders | interventions — Genetic Counseling

STUDY DESIGN:
Intervention Model Description: Trial-within-cohort
Who Masked: Outcomes Assessor
Masking Description: Eligible participants who are randomized to not be offered the intervention will not be aware of the presence of a potential intervention. Study staff who are assessing outcomes (i.e., psychopathology, cannabis use) will not know who did and did not receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Genetic counselling (Experimental): Eligible participants who are randomized will be contacted and offered an invitation to attend the intervention. Genetic counselling will be provided to participants who accept the intervention as a single 1-2 hour session by a board-certified genetic counsellor. During the genetic counselling session, participants will have the option to receive their genotype at rs2494732. Participants will be counselled regarding their individualized risk of developing and of NOT developing SMI based on family history, whether or not they choose to use cannabis, and genotype (if they accept the genetic test results). Approximately 1 month after the intervention, participants will receive a follow-up interview.
  Interventions: Behavioral: Genetic counselling
- Control group (No Intervention): Eligible participants who are not randomized to be offered the intervention will continue with their annual assessments as part of the parent study. These participants will receive the current standard of care (no intervention), and will not be offered or informed of the intervention.

INTERVENTIONS:
Behavioral: Genetic counselling — Participants will receive information on risk/protective factors and causes of mental illness. Participants are not required to receive numeric/genetic risk information. Participants who choose to receive genetic and/or numeric risk information will be counselled on their risk of NOT developing and of developing SMI based on their genetic test results and/or family history information they provide. Risk estimates will be derived by genetic counsellors, according to standard practice guidelines. Participants who receive genetic information will be counselled on the possible influence of cannabis use on risk of mental illness based on their genotype. Participants who choose to not receive genetic information will be counselled on the influence of cannabis on mental health.
  Arms: Genetic counselling

SUMMARY:
Severe mental illness (SMI) refers to the most burdensome psychiatric conditions. The need to pre-empt the onset of SMI is pressing because once SMI develops, quality of life is poor and available treatments have limited efficacy. Most risk factors for SMI are either unchangeable (e.g., genetics) or difficult to alter (e.g., low socio-economic status). In contrast, cannabis use is one specific risk factor that could be avoided. Certain individuals are more vulnerable to the harmful effects of cannabis. Genetic factors can help us identify these high-risk individuals. One in three individuals are carriers of a higher-risk genetic variant, and cannabis users with this genotype are at up to 7-fold increased risk of developing schizophrenia. In our study, genetic counselling will be provided to participants by a board-certified genetic counsellor. During the genetic counselling session, participants will have the option to receive their genotype. Participants will be counselled regarding their individualized risk of developing and of not developing SMI based on family history, whether or not they choose to use cannabis, and genotype (if the participants accept the genetic test results). The investigators hypothesize that this intervention will reduce exposure to cannabis compared to the youth who are not offered the intervention.

DETAILED DESCRIPTION:
Severe mental illness (SMI) refers to the most burdensome forms of psychiatric disorder, including schizophrenia, bipolar disorder, and severe depression. These illnesses typically emerge in adolescence or young adulthood and are associated with substantial impairment in functioning. A significant proportion (~30%) of individuals with SMI remain resistant to any form of available pharmacotherapy. The combination of early onset, poor response to treatment and persistent disability makes SMI the most problematic group of illnesses to individuals and society. The need for early interventions to pre-empt the onset of SMI is pressing because once SMI develops, quality of life is poor for patients and their families. There is substantial overlap in the genetic and environmental risk factors for individual forms of SMI, and predictors of SMI are not specific to any one disorder. It is therefore necessary to conceptualize SMI as transdiagnostic and include diagnoses of schizophrenia, bipolar disorder, and depression, rather than focusing on single illnesses when developing preventative interventions. Prevention of SMI is currently hindered by the inability to identify those at risk early enough to normalize their developmental trajectory. Recent advances in genomics and the understanding of important gene-environment interactions may help overcome this challenge and enable effective and targeted prevention of SMI. Cannabis exposure during critical periods of brain maturation is an avoidable environmental risk factor for SMI. A replicated gene-cannabis interaction shows that carriers of a common genetic variant (C alleles at rs2494732 in the AKT1 gene) are at up to 7-fold increased risk of developing psychosis if they use cannabis. Genetic counselling provides a powerful tool to communicate genetic information to youth in a way that empowers and enhances health. The present project involves the delivery of a genetic counselling intervention to inform youth of their personalized risk of developing SMI based on genotype, family history, and whether or not they choose to use cannabis. This project will be the first application of molecular genetic information and genetic counselling to prevent SMI.

Aim: To test if genetic counselling regarding personalized risk information based on a replicated gene-cannabis interaction reduces cannabis use in youth at high risk of developing severe mental illness.

Hypotheses:

1. A genetic counselling intervention will be acceptable to youth at high familial risk of SMI.
2. A genetic counselling intervention with personalized feedback of AKT1 genotype will reduce cannabis use among vulnerable youth.
3. The effect of the intervention will be moderated by AKT1 genotype, with greater reduction of cannabis use among carriers of the sensitive C alleles.

Method: A cohort of over 450 youth (aged 3-29) has been enrolled as part of the Families Overcoming Risks and Building Opportunities for Well-being (FORBOW) study. The investigators have obtained biological samples for measurement of genetic variation and the investigators will obtain biological samples to measure cannabis exposure. The investigators will randomly select one in every two eligible youth (aged 12-21) to be offered genetic counselling during which the participants will be provided with personalized genetic information and they will be counselled regarding risk of developing SMI based on genotype, family history, and whether or not they choose to use cannabis. The investigators will follow the participants through the developmental period with the highest risk of cannabis use initiation and the investigators will assess cannabis use and psychopathology annually. The primary outcome will be abstinence from cannabis reported by participants in confidential interviews and confirmed by measurement of the primary metabolites of psychoactive Δ9-tetrahydrocannabinol in blood and urine samples.

Significance: This project will realize the first translational application of a gene-environment interaction to improve mental health and test an intervention with potential public health benefits.

ELIGIBILITY:
Inclusion Criteria:

* Enrolment in the Families Overcoming Risks and Building Opportunities for Well-being (FORBOW) study.
* Age between 12 and 21 years.
* Knowledge of English sufficient to benefit from the intervention.
* Capacity to provide informed consent at most recent FORBOW assessment.
* Provision of consent to be contacted about future studies at most recent FORBOW assessment.

Exclusion Criteria:

* A diagnosis of severe mental illness (psychotic disorder, bipolar disorder, severe/recurrent depression) at baseline
* Autism or intellectual disability of a degree that interferes with assessment (IQ < 70)

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported cannabis use | 1 month
  Self-reported cannabis use on a questionnaire.

SECONDARY OUTCOMES:
The proportion of participants who complete the intervention after receiving an offer to participate (intervention acceptability) | Completion of study (2 years).
  Acceptability will be established as the proportion of individuals accepting the offer of intervention.
Presence of cannabinoids in urine | 1 month
  Urine will be screened for the presence/absence of cannabinoids.

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Uher, MD, PhD, Principal Investigator — Nova Scotia Health Authority, Dalhousie University
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zwicker A, LeBlanc MA, Pavlova B, Alda M, Denovan-Wright EM, Uher R, Austin JC. Genetic counselling for the prevention of mental health consequences of cannabis use: A randomized controlled trial-within-cohort. Early Interv Psychiatry. 2021 Oct;15(5):1306-1314. doi: 10.1111/eip.13082. Epub 2020 Nov 26. PMID 33242924
- See also: FORBOW study website. — http://www.forbow.org